CLINICAL TRIAL: NCT04188834
Title: Neurophysiological and Behavioral Effects of Sensory Flicker and Electrical Flicker Stimulation
Brief Title: Effects of Sensory Flicker and Electrical Flicker Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, Joseph R Manns, PhD, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00107577
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-02

CONDITIONS: Brain Diseases
Keywords: Sensory Flicker Stimulation; Electrical Flicker Stimulation; Neurophysiological Effects; Behavioral Effects; Brain circuits modulation; Steady-state evoked potentials
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sensory Flicker Stimulation (Experimental): Participants will be exposed for about 10 to 60 minutes at a time, to a sequence of sensory flicker trials each lasting a few seconds to 5 minutes, while their eyes are open or closed. Each trial may include the following modalities and frequencies of flicker:
  * Modalities: auditory only, visual only, or audiovisual combined.
  * Frequencies: random, or anywhere from 3Hz to 200Hz.
  Additionally, subjects may be exposed to individual pulses of light and/or sound, i.e. around or less than 1 pulse /second, for up to 20 minutes at a time.
  Interventions: Device: Customized version of DAVID device
- Electrical Flicker Stimulation (Active Comparator): Participants will be exposed to direct electrical brain stimulation with low-amplitude current, at given flicker frequencies. Participants will be exposed to frequencies ranging from 5-100Hz, for up to 10 seconds at a time. Initially, frequencies of 5.5Hz and 40Hz will be tested.
  During brain stimulation sessions, bipolar electrical stimulation will be applied to one or more areas of the brain at a time either with or without associated memory tasks. Stimulation in the absence of any memory task will be applied to assess the subject's neurophysiological response to stimulation and to identify the optimal stimulation parameters for use during memory tasks. Stimulation during behavioral tasks will be applied in an attempt to affect the subject's memory.
  Interventions: Device: Blackrock CereStim

INTERVENTIONS:
Device: Customized version of DAVID device — A customized version of the DAVID device will be used to expose participants to sensory flicker. The device consists of opaque glasses containing LEDs to present flickering light, as well as earbuds or headphones to present flickering sound.
  Arms: Sensory Flicker Stimulation
Device: Blackrock CereStim — The Blackrock CereStim is a fully programmable neurostimulator. The current pulses generated by the Blackrock CereStim are intended to stimulate neurons in proximity to a set of electrodes.
  Arms: Electrical Flicker Stimulation

SUMMARY:
The study will evaluate whether sensory flicker can modulate neural activity of deep brain regions in humans, and whether it can have relevant effects on behavior. Moreover, it will compare those effects to the gold-standard method of modulating brain circuits, direct electrical stimulation of the brain (the same mechanism as deep brain stimulation), using a powerful within-subjects design.

DETAILED DESCRIPTION:
Clinical trials have explored the modulation of brain circuits to treat several brain disorders, including Parkinson's Disease, Alzheimer's Disease (AD), depression, and Obsessive-Compulsive Disorder (OCD). However, current means to non-invasively modulate brain activity are limited.

The study will evaluate whether sensory flicker can modulate neural activity of deep brain regions in humans, and whether it can have relevant effects on behavior. Moreover, it will compare those effects to the gold-standard method of modulating brain circuits, direct electrical stimulation of the brain (the same mechanism as deep brain stimulation), using a powerful within-subjects design.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years, regardless of gender, race or ethnicity).
* To be implanted with intracranial depth or grid/strip electrodes for surgical evaluation.
* Patient was not shown, during phase I seizure monitoring, to exhibit abnormal EEG activity in response to photic stimulation, and is not clinically suspected to be susceptible to photic-induced seizures.
* Patient has no pre-existing diagnosis of autism.
* Patient is not considered at risk for psychogenic nonepileptic seizures (PNES) triggered by sensory stimulation.
* Fluent in English.
* Able to understand an informed consent (comprehend potential risks and benefits).
* Give written and verbal informed consent to all experiments patient would participate in.

Exclusion Criteria:

* Failure to meet any one inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Manns, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant and data that underlie the results reported after de-identification (text, tables, figures, and appendices) will be available. The study protocol, statistical analysis plan, analytic code will be made available immediately following publication with no end date.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: De-identified, minimally processed data and processed data will be made available upon request. Data may be requested by contacting Dr. Annabelle Singer at annabelle.singer@bme.edu

REFERENCES:
- [Background] Blanpain LT, Chen E, Park J, Walelign MY, Gross RE, Cabaniss BT, Willie JT, Singer AC. Multisensory Flicker Modulates Widespread Brain Networks and Reduces Interictal Epileptiform Discharges in Humans. medRxiv [Preprint]. 2023 Mar 17:2023.03.14.23286691. doi: 10.1101/2023.03.14.23286691. PMID 36993248
- See also: Multisensory Flicker Modulates Widespread Brain Networks and Reduces Interictal Epileptiform Discharges in Humans — https://pubmed.ncbi.nlm.nih.gov/36993248/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory University Hospital in Atlanta, Georgia, USA. Participant enrollment began January 10, 2020, and all follow up was complete by November 22, 2022.
Pre-assignment Details: Participants only had the Sensory Flicker Stimulation. In the initial IRB protocol submission, the research team intended to potentially do electrical flicker experiments as further exploration of their project but ended up opting not to pursue this avenue.
Groups:
- Sensory Flicker Stimulation: Participants will be exposed for about 10 to 60 minutes at a time, to a sequence of sensory flicker trials each lasting a few seconds to 5 minutes, while their eyes are open or closed. Each trial may include the following modalities and frequencies of flicker:
  * Modalities: auditory only, visual only, or audiovisual combined.
  * Frequencies: random, or anywhere from 3Hz to 200Hz.
  Additionally, subjects may be exposed to individual pulses of light and/or sound, i.e. around or less than 1 pulse /second, for up to 20 minutes at a time.
  Customized version of DAVID device: A customized version of the DAVID device will be used to expose participants to sensory flicker. The device consists of opaque glasses containing LEDs to present flickering light, as well as earbuds or headphones to present flickering sound.
Period: Overall Study
Arm/Group | Sensory Flicker Stimulation
Started | 23
Completed | 19
Not Completed | 4
Not completed — Participants did not complete enough proportion of experiment(s) to be included in analysis | 4

BASELINE CHARACTERISTICS:
Arm/Group | Sensory Flicker Stimulation
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Fold-change in Oscillatory Activity (Power Spectral Density) in Response to Exposure to Sensory Flicker: Comparing Mean Power Spectral Density at the Frequency of Flicker Being Presented Between Flicker and Baseline Periods
Description: The power spectral density of the LFP will be measured across stimulus frequencies and modalities of sensory flicker stimuli in visual areas, auditory areas, hippocampus, and prefrontal cortex. To evaluate the effects of sensory flicker on brain activity in various brain regions, researchers compared the average increase in oscillatory neural activity of given recorded brain regions during sensory stimulation, among the total number of recording locations that showed a significant response to sensory stimulation compared to baseline. In participants in whom a condition was repeated across multiple experimental sessions. If a location showed a significant response in multiple sessions, the data point that showed the highest level of response was kept. The average fold-change increase in oscillatory activity, 25th and 75th percentiles, within a region of interest is reported.
Time Frame: During experiment session (up to 2 hours) during hospital admission (up to 2 weeks)
Population: Participants who completed study procedures and had valid data points for each frequency and region are included.
Measure: Median (Inter-Quartile Range); unit: Fold-change in power
Arm/Group | Sensory Flicker Stimulation
Number analyzed (Participants) | 19
Fold-change in power
  Visual Region to 5.5Hz-V: number analyzed (Participants) | 8
  Visual Region to 5.5Hz-V | 4.6 [1.2 to 11.2]
  Visual Region to 40Hz-V: number analyzed (Participants) | 8
  Visual Region to 40Hz-V | 4 [1.3 to 15.8]
  Visual Region to 80Hz-V: number analyzed (Participants) | 8
  Visual Region to 80Hz-V | 1.1 [0.6 to 3.5]
  Visual Region to 5.5Hz-A: number analyzed (Participants) | 7
  Visual Region to 5.5Hz-A | 0.5 [0.4 to 0.7]
  Visual Region to 40Hz-A: number analyzed (Participants) | 7
  Visual Region to 40Hz-A | 0.4 [0.3 to 0.8]
  Visual Region to 80Hz-A: number analyzed (Participants) | 7
  Visual Region to 80Hz-A | 0.6 [0.4 to 0.7]
  Auditory Region to 5.5Hz-V: number analyzed (Participants) | 15
  Auditory Region to 5.5Hz-V | 0.9 [0.6 to 2.0]
  Auditory Region to 40Hz-V: number analyzed (Participants) | 15
  Auditory Region to 40Hz-V | 0.7 [0.5 to 3.5]
  Auditory Region to 80Hz-V: number analyzed (Participants) | 15
  Auditory Region to 80Hz-V | 0.7 [0.4 to 3.6]
  Auditory Region to 5.5Hz-A: number analyzed (Participants) | 16
  Auditory Region to 5.5Hz-A | 0.7 [0.5 to 1.2]
  Auditory Region to 40Hz-A: number analyzed (Participants) | 16
  Auditory Region to 40Hz-A | 1.6 [0.6 to 4.6]
  Auditory Region to 80Hz-A: number analyzed (Participants) | 16
  Auditory Region to 80Hz-A | 1 [0.5 to 3.4]
  Medial temporal lobe (MTL) Region to 5.5Hz-V: number analyzed (Participants) | 15
  Medial temporal lobe (MTL) Region to 5.5Hz-V | 0.6 [0.5 to 1.4]
  MTL Region to 40Hz-V: number analyzed (Participants) | 15
  MTL Region to 40Hz-V | 0.8 [0.5 to 1.4]
  MTL Region to 80Hz-V: number analyzed (Participants) | 15
  MTL Region to 80Hz-V | 0.6 [0.4 to 0.9]
  MTL Region to 5.5Hz-A: number analyzed (Participants) | 16
  MTL Region to 5.5Hz-A | 0.7 [0.5 to 1.6]
  MTL Region to 40Hz-A: number analyzed (Participants) | 16
  MTL Region to 40Hz-A | 0.6 [0.4 to 1.1]
  MTL Region to 80Hz-A: number analyzed (Participants) | 16
  MTL Region to 80Hz-A | 0.5 [0.4 to 0.6]
  PFC Region to 5.5Hz-V: number analyzed (Participants) | 12
  PFC Region to 5.5Hz-V | 0.5 [0.4 to 0.9]
  PFC Region to 40Hz-V: number analyzed (Participants) | 12
  PFC Region to 40Hz-V | 0.5 [0.4 to 1]
  PFC Region to 80Hz-V: number analyzed (Participants) | 12
  PFC Region to 80Hz-V | 0.5 [0.4 to 1.2]
  PFC Region to 5.5Hz-A: number analyzed (Participants) | 14
  PFC Region to 5.5Hz-A | 0.5 [0.4 to 0.6]
  PFC Region to 40Hz-A: number analyzed (Participants) | 14
  PFC Region to 40Hz-A | 0.5 [0.4 to 0.5]
  PFC Region to 80Hz-A: number analyzed (Participants) | 14
  PFC Region to 80Hz-A | 0.4 [0.3 to 0.6]

2. Secondary Outcome: Effect of Sensory Flicker on the Rate of Interictal Epileptiform Discharges (IEDs) Which Represent Pathological Activity Often Observed in Epilepsy
Description: The change of of the sensory flicker effect will be evaluated by the comparison of the whole-brain rate of IEDs between sensory flicker stimulation and baseline (no stimulation).
Time Frame: During experiment session (up to 2 hours) during hospital admission (up to 2 weeks)
Population: Participants who completed study procedures and had valid data points for each frequency and region are included.
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Sensory Flicker Stimulation
Number analyzed (Participants) | 19
Percent change | -3.0 [-4.5 to -1.6]

ADVERSE EVENTS:
Time Frame: Adverse events that occurred during the experimental sessions (up to 2h) and were conducted during the patient's hospital stay are reported. Participant's hospital stay duration was strictly determined by the clinical team based on clinical needs and typically lasted about 2 weeks.
Arm/Group | Sensory Flicker Stimulation
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 16/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensory Flicker Stimulation (N=23)
Headache or discomfort (Nervous system disorders) | 8 (10)
Fatigue (General disorders) | 8 (10)
Miscellaneous (General disorders) | 8 (8)
Seizure likely unrelated to experiment (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT04188834/Prot_SAP_001.pdf